CLINICAL TRIAL: NCT03512652
Title: Clinical Study to Assess the Effectiveness of the Device Patello
Acronym: Patello
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SUPSI
Record Dates: First submitted 2018-04-03; First posted 2018-05-01 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Passiv Continuous Patella Mobilisation

STUDY DESIGN:
Intervention Model Description: The right knee is treated by the intervention device Patello
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patello (Experimental): The participants' right knee was placed inside the patello device, a total of 50 repetitions, with a constant mobilisation speed, was conducted and the degree of translation was assessed after 1, 10, 20, 30 and 50 repetitions.
  Interventions: Device: Patello

INTERVENTIONS:
Device: Patello — The Patello is a new intervention device which mobilizes the Patella passively and continuously in cranial-caudal direction to increase Patella mobility.

SUMMARY:
The device "Patello" was designed to passively mobilize the Patella in cranial-caudal direction. Its application field lays in the rehabilitation of any knee pathology where knee range of motion may be restricted due to the Patella mobility.

DETAILED DESCRIPTION:
The effectiveness of the device Patello has not been tested so far. This clinical study aims to assess and proof the effectiveness of this device. The aim is to objectify the movement of the Patella induced by the device Patello in cranial / caudal direction. As outcome parameter serve ultrasound measurements of a bony reference point of the femur and the Patella and its displacement / distance after mobilization.

ELIGIBILITY:
Inclusion Criteria:

* no operation and / or actual problems (pain at rest or during strain) of the muscular or bony parts of the lower extremities
* closed and intact skin conditions in the area of the knees and thighs
* no fear of the intervention
* willingness to participate on all 2 measurement days

Exclusion Criteria:

* operation and / or actual problems (pain at rest or during strain) of the muscular or bony parts of the lower extremities
* open skin conditions in the area of the knees and thighs
* fear of the intervention
* no willingness to participate on all 2 measurement days

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, Dr, Principal Investigator — University of Applied Sciences and Art of Switzerland (SUPSI)
Locations (1):
- SUPSI Landquart, Landquart, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hohenauer, E., Stoop, R., Koller, A., Gredig, J., Fenzl, M., Deflorin, C., & Clijsen, R. (2020). Efficacy of a new device for passive continuous patellar mobilization. International Journal of Medical and Biomedical Studies, 4(3), 07-10. doi: 10.32553/ijmbs.v4i3.971
- See also: fullversion of publication — https://ijmbs.info/index.php/ijmbs/article/view/971
- Available data/document: scientific Article — https://ijmbs.info/index.php/ijmbs/article/view/971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patello
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patello
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  Switzerland | 9

OUTCOME MEASURES:

1. Primary Outcome: Patellofemoral Translation
Description: Patellar cranial-caudal translation (in centimeters) is assessed repeatedly within a single passive continuous mobilization session. A total of 50 repetitions are performed at a constant mobilization speed. Ultrasound video sequences are recorded, and patellar translation is analyzed immediately after 1, 10, 20, 30, and 50 repetitions during the same session.
Time Frame: Assessed after 1, 10, 20, 30 and 50 mobilization repetitions during a single continous passieve patellar moblizitaion session of 50 repetitions (total duration approximately 5-10 minutes)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Patello
Number analyzed (Participants) | 9
cm
  1 repetition | 0.819 (0.396)
  10 repetitions | 0.734 (0.280)
  20 repetitions | 0.776 (0.307)
  30 rep. | 0.771 (0.300)
  50 rep. | 0.774 (0.297)

ADVERSE EVENTS:
Time Frame: Immediate duration of the intervention session (up to 50 repetitions), around 70 minutes
Arm/Group | Patello
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03512652/Prot_SAP_000.pdf